CLINICAL TRIAL: NCT03307590
Title: Adding Dexmedetomidine to Caudal Bupivacaine for Analgesia in Supra - Umbilical Pediatric Surgeries: Would it Add More Analgesia
Brief Title: Comparing Dexmedetomidine With Bupivacaine Versus Bupivacaine Alone for Caudal Block in Supra - Umbilical Surgeries
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Kareem, Anesthesiologist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Caudaldexsupraumblical
Record Dates: First submitted 2017-08-20; First posted 2017-10-11 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Anesthesia
MeSH Terms: interventions — Dexmedetomidine; Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- D group (Active Comparator): Dexmedetomidine with bupivacaine group Caudal dexmedetomidine 1.5 microgram/kg with bupivavaine (0.25%) 1.25 ml/kg were administered
  Interventions: Drug: Dexmedetomidine
- B group (Active Comparator): Bupivacaine only group Caudal bupivavaine (0.25%) 1.25 ml/kg without dexmedetomidine was administered
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Dexmedetomidine — Caudal block by dexmedetomidine and bupivavaine
  Other Names: Precedex
  Arms: D group
Drug: Bupivacaine — Caudal block by bupivavaine alone
  Other Names: Marcaine
  Arms: B group

SUMMARY:
dexmedetomidine is an alpha 2 adrenergic receptor agonist that is given either systemically or combined to local anesthetics during regional blocks. Investigators studied the combination of dexmedetomedine/bupivacaine versus bupivacaine alone for caudal blockage in pediatric patients undergoing supra - umbilical surgeries.

DETAILED DESCRIPTION:
Dexmedetomidine was combined to bupivavaine and administered via caudal route to be compared to caudal bupivavaine alone for analgesia following upper trunk surgery

ELIGIBILITY:
Inclusion Criteria:

* supra - umbilical surgeries

Exclusion Criteria:

* allergy to the drug or coagulopathy

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Pain relief | 6 months study
  CHEOPS scale value

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided